CLINICAL TRIAL: NCT00197002
Title: A Phase IIIb, Open, Randomized, Controlled, Multicenter Study of the Immunogenicity and Safety of GSK Biologicals' Inactivated Hepatitis A Vaccine Administered on a 0-6 Mth Schedule Concomitantly With Wyeth Lederle's Pneumococcal Conjugate Vaccine in Healthy Children 15 Months of Age
Brief Title: Immune Response & Safety of a Hepatitis A Vaccine Given Together With a Pneumococcal Vaccine in Healthy Children 15 m of Age
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 208109/220
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Results first posted 2017-02-20 (Actual); Last update posted 2018-08-06 (Actual); Status verified 2018-06

CONDITIONS: Hepatitis A
MeSH Terms: conditions — Hepatitis A | interventions — Hepatitis A Vaccines; Heptavalent Pneumococcal Conjugate Vaccine

ARMS (3):
- Havrix Group (Active Comparator): Healthy male or female subjects, 15 months of age, who received Havrix® vaccine administered intramuscularly in the right anterolateral thigh, at Day 0 and at Month 6-9.
  Interventions: Biological: GSK Biologicals 2-dose inactivated hepatitis A vaccine (Havrix)
- Havrix+Prevnar Group (Experimental): Healthy male or female subjects, 15 months of age, who received Havrix® and Prevnar™ vaccines co-administered intramuscularly in the right and left anterolateral thighs, respectively, at Day 0 and Havrix® vaccine administered intramuscularly in the right anterolateral thigh, at Month 6-9.
  Interventions: Biological: GSK Biologicals 2-dose inactivated hepatitis A vaccine (Havrix); Biological: Prevnar™
- Prevnar Havrix Group (Active Comparator): Healthy male or female subjects, 15 months of age, who received Prevnar™ vaccine administered intramuscularly in the left anterolateral thigh, at Day 0 and Havrix® vaccine, administered intramuscularly in the right anterolateral thigh, at Day 30 and at Month 7-10.
  Interventions: Biological: GSK Biologicals 2-dose inactivated hepatitis A vaccine (Havrix); Biological: Prevnar™

INTERVENTIONS:
Biological: GSK Biologicals 2-dose inactivated hepatitis A vaccine (Havrix) — Two doses, administered intramuscularly in the right anterolateral thigh.
Biological: Prevnar™ — One dose, administered intramuscularly in the left anterolateral thigh.
  Arms: Havrix+Prevnar Group; Prevnar Havrix Group

SUMMARY:
This is a study to evaluate the immunogenicity and safety of GSK Biologicals 2-dose inactivated hepatitis A vaccine when administered with a pneumococcal conjugate vaccine in children as young as 15 months of age.

DETAILED DESCRIPTION:
An open, controlled comparison of Havrix administered alone or with Prevnar. The three groups evaluated are: 1) Havrix alone, 2) Havrix plus Prevnar and 3) Prevnar followed by Havrix one month later.

ELIGIBILITY:
Inclusion Criteria:

* A male or female child 12 or 13 months of age at the time of entry into the Enrollment Phase,
* Free of obvious health problems,
* Subjects must have previously received three doses of Prevnar in his/her first year of life.

Exclusion Criteria:

* Use of any investigational or non-registered drug or vaccine within 42 days preceding the first dose of study vaccine, or planned use during the study period,
* Chronic administration of immuno-suppressant or other immune-modifying drugs within six months prior to vaccination or planned administration at any time during the study period. (For corticosteroids, this will mean prednisone, or equivalent, less than 0.5 mg/kg/day. Inhaled, nasal and topical steroids are allowed.),
* Administration of the ACIP-recommended fourth dose of Prevnar prior to entering the Enrollment Phase of the study,
* Planned administration or administration of any vaccine not foreseen by the study protocol within the period of 42 days before and 30 days after each dose of study vaccine(s),
* Previous vaccination against hepatitis A,
* History of hepatitis A or known exposure to hepatitis A,
* Any confirmed or suspected immunosuppressive or immunodeficient condition, including human immunodeficiency virus (HIV) infection,
* A family history of congenital, hereditary or infectious immunodeficiency or parental risk factors for HIV infection,
* History of allergic disease/reactions or hypersensitivity likely to be exacerbated by any component of Havrix (e.g., neomycin, 2-phenoxyethanol) or Prevnar (e.g., diphtheria toxoid),
* Major congenital defects or serious chronic illness,
* History of any neurologic disorder (history of febrile seizures not associated with an underlying neurological disorder does not exclude the subject),
* Acute disease, defined as the presence of a moderate or severe illness with or without fever, at the time of vaccination,
* Administration of immunoglobulins and/or any blood products within three months prior to the first dose of study vaccine or planned administration at any time during the entire study period.

Ages: 12 Months to 13 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 521 (Actual)
Dates: Start 2003-09-11 (Actual); Primary Completion 2006-01-16 (Actual); Study Completion 2006-01-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (16):
- United States (16):
  - GSK Investigational Site, Centennial, Colorado
  - GSK Investigational Site, Bardstown, Kentucky
  - GSK Investigational Site, Louisville, Kentucky
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Kalamazoo, Michigan
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, North Las Vegas, Nevada
  - GSK Investigational Site, Stony Brook, New York
  - GSK Investigational Site, Chapel Hill, North Carolina
  - GSK Investigational Site, University Heights, Ohio
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Salt Lake City, Utah
  - GSK Investigational Site, Vancouver, Washington

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Trofa AF, Levin M, Marchant CD, Hedrick J, Blatter MM. Immunogenicity and safety of an inactivated hepatitis a vaccine administered concomitantly with a pneumococcal conjugate vaccine in healthy children 15 months of age. Pediatr Infect Dis J. 2008 Jul;27(7):658-60. doi: 10.1097/INF.0b013e31816907bd. PMID 18536623
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: 208109/220 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 208109/220 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 208109/220 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 208109/220 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 208109/220 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 208109/220 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Out of a total of 521 subjects enrolled, 88 subjects were not administered a study vaccine dose and thus were not considered to have started the study.
Period: Overall Study
Arm/Group | Havrix Group | Havrix+Prevnar Group | Prevnar Havrix Group
Started | 147 | 137 | 149
Completed | 125 | 119 | 132
Not Completed | 22 | 18 | 17
Not completed — Adverse Event | 0 | 1 | 0
Not completed — Protocol Violation | 1 | 0 | 2
Not completed — Withdrawal by Subject | 9 | 5 | 7
Not completed — Migrated/moved from study area | 3 | 5 | 1
Not completed — Lost to follow-up (incompl. vaccination) | 4 | 4 | 5
Not completed — Lost to follow-up (compl. vaccination) | 2 | 2 | 1
Not completed — Others | 3 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Havrix Group | Havrix+Prevnar Group | Prevnar Havrix Group | Total
Number analyzed (Participants) | 147 | 137 | 149 | 433
Age, Continuous [Mean (Standard Deviation); unit: Months] | 15.0 (0.16) | 15.0 (0.09) | 15.0 (0.24) | 15.0 (0.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 77 | 66 | 79 | 222
  Male | 70 | 71 | 70 | 211

OUTCOME MEASURES:

1. Primary Outcome: Number of Seropositive Subjects for Anti-HAV Antibodies
Description: Cut-off values assessed were greater than or equal to (≥) 15 milli-international units per milliliter (mIU/mL) in the sera of subjects seronegative before vaccination.
Time Frame: At one month after Dose 2 of Havrix® vaccine (Month 7-10)
Population: The analysis was performed on the According-to-Protocol (ATP) cohort for immunogenicity, which included all vaccinated subjects for whom immunogenicity data were available and who complied with the eligibility criteria as defined in the protocol.
Measure: Count of Participants; unit: Participants
Arm/Group | Havrix Group | Havrix+Prevnar Group
Number analyzed (Participants) | 106 | 94
Participants | 106 | 94
Statistical Analysis 1: Comparison: Havrix Group vs Havrix+Prevnar Group; Difference in seropositivity rates for anti-HAV: To demonstrate the non-inferiority of Havrix® vaccine co-administered with Prevnar™ vaccine (Havrix+Prevnar Group), compared to Havrix® vaccine administered alone (Havrix Group), in terms of seropositivity rates and geometric mean concentrations (GMCs) for anti-HAV antibody, one month after Dose 2 of Havrix® vaccine (Month 7-10); Test type: Non-Inferiority or Equivalence — The two-sided standardized asymptotic 95% confidence interval (CI) for the difference in seropositivity rates [Havrix+Prevnar Group minus Havrix Group] was computed. The anti-HAV seropositivity rates in the Havrix+Prevnar Group were considered as non-inferior to the seropositivity rates in the Havrix Group, if the lower limit of the 95% CI was not lower (≥) than -5%. The non-inferiority was concluded if both non-inferiority criteria (for seropositivity rates and GMCs) were met; Difference in seropositivity rate = -1.06, 95% CI 2-sided [-5.78 to 2.45]

2. Primary Outcome: Concentrations for Anti-HAV Antibodies
Description: Anti-HAV antibody concentrations are presented as geometric mean concentrations (GMCs), expressed in milli-international units per milliliter (mIU/mL).
Time Frame: At one month after Dose 2 of Havrix® vaccine (Month 7-10)
Population: The analysis was performed on the ATP cohort for immunogenicity, which included all vaccinated subjects for whom immunogenicity data were available and who complied with the eligibility criteria as defined in the protocol.
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Havrix Group | Havrix+Prevnar Group
Number analyzed (Participants) | 106 | 94
mIU/mL | 1609.9 [1254.9 to 2065.3] | 1526.4 [1196.2 to 1947.8]
Statistical Analysis 1: Comparison: Havrix Group vs Havrix+Prevnar Group; To demonstrate the non-inferiority of Havrix® vaccine co-administered with Prevnar™ vaccine (Havrix+Prevnar Group), compared to Havrix® vaccine administered alone (Havrix Group), in terms of seropositivity rates and geometric mean concentrations (GMCs) for anti-HAV antibody, one month after Dose 2 of Havrix® vaccine (Month 7-10); Test type: Non-Inferiority or Equivalence — The standardized two-sided 95% CI for the GMC ratio (Havrix+Prevnar Group divided by Havrix Group) was computed. The anti-HAV GMC in the Havrix+Prevnar Group was considered as non-inferior to the anti-HAV GMC in the Havrix Group if the lower limit of the 95% CI was not lower than (≥) 0.5. The non-inferiority of the anti-HAV immune response in Havrix+Prevnar Group compared to Havrix Group was concluded if both non-inferiority criteria (for seropositivity rates and GMCs) were met; ANCOVA; Adjusted GMC ratio = 0.91, 95% CI 2-sided [0.63 to 1.31]

3. Secondary Outcome: Anti-4, Anti-6B, Anti-9V, Anti-14, Anti-19F and Anti-23F Antibody Concentrations
Description: Antibody concentrations against pneumococcal serotypes (4, 6B, 9V, 14, 18C, 19F and 23F) are presented as geometric mean concentrations (GMCs), expressed in microgram per milliliter (μg/mL).
Time Frame: At one month after Prevnar™ vaccination (Day 30)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Havrix+Prevnar Group | Prevnar Havrix Group
Number analyzed (Participants) | 102 | 117
μg/mL
  Anti-4: number analyzed (Participants) | 102 | 115
  Anti-4 | 3.3 [2.8 to 3.9] | 3.1 [2.6 to 3.7]
  Anti-6B: number analyzed (Participants) | 101 | 117
  Anti-6B | 7.1 [5.8 to 8.6] | 6.1 [4.8 to 7.6]
  Anti-9V: number analyzed (Participants) | 101 | 116
  Anti-9V | 6.8 [5.8 to 7.9] | 7.4 [6.3 to 8.8]
  Anti-14: number analyzed (Participants) | 101 | 116
  Anti-14 | 9.8 [8.3 to 11.7] | 11.2 [9.5 to 13.2]
  Anti-18C: number analyzed (Participants) | 101 | 115
  Anti-18C | 5.8 [5.0 to 6.8] | 5.7 [4.7 to 7.0]
  Anti-19F: number analyzed (Participants) | 101 | 116
  Anti-19F | 2.8 [2.3 to 3.2] | 2.6 [2.2 to 3.1]
  Anti-23F: number analyzed (Participants) | 101 | 116
  Anti-23F | 9.0 [7.4 to 11.0] | 7.9 [6.4 to 9.7]

4. Secondary Outcome: Number of Subjects With an Immune Response to Anti-pneumococcal Serotypes 4, 6B, 9V, 14, 18C, 19F and 23F
Description: The immune response was defined, with respect to anti-pneumococcal response rates, as an antibody concentration equal to or above (≥) 0.05 μg/mL.
Time Frame: At one month after Prevnar™ vaccination (Day 30)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Havrix+Prevnar Group | Prevnar Havrix Group
Number analyzed (Participants) | 102 | 117
Participants
  Anti-4: number analyzed (Participants) | 102 | 115
  Anti-4 | 102 | 115
  Anti-6B: number analyzed (Participants) | 101 | 117
  Anti-6B | 100 | 115
  Anti-9V: number analyzed (Participants) | 101 | 116
  Anti-9V | 101 | 116
  Anti-14: number analyzed (Participants) | 101 | 116
  Anti-14 | 101 | 116
  Anti-18C: number analyzed (Participants) | 101 | 115
  Anti-18C | 101 | 114
  Anti-19F: number analyzed (Participants) | 101 | 116
  Anti-19F | 101 | 116
  Anti-23F: number analyzed (Participants) | 101 | 116
  Anti-23F | 100 | 115

5. Secondary Outcome: Number of Seropositive Subjects for Anti-HAV Antibodies
Description: Cut-off values assessed were greater than or equal to (≥) 15 mIU/mL in the sera of subjects seronegative before vaccination.
Time Frame: At one month after Dose 1 of Havrix® vaccine (Day 30)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Havrix Group | Havrix+Prevnar Group
Number analyzed (Participants) | 119 | 103
Participants | 100 | 91

6. Secondary Outcome: Concentrations for Anti-HAV Antibodies
Description: Anti-HAV antibody concentrations are presented as geometric mean concentrations (GMCs), expressed in milli international units per milliliter (mIU/mL).
Time Frame: At one month after Dose 1 of Havrix® vaccine (Day 30)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Havrix Group | Havrix+Prevnar Group
Number analyzed (Participants) | 119 | 103
mIU/mL | 48.0 [39.4 to 58.5] | 61.0 [49.3 to 75.4]

7. Secondary Outcome: Number of Seropositive Subjects for Anti-HAV Antibodies
Description: as for outcome 5
Time Frame: At one month after Dose 2 of Havrix® vaccine (Month 8-11)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Prevnar Havrix Group
Number analyzed (Participants) | 115
Participants | 113

8. Secondary Outcome: Concentrations for Anti-HAV Antibodies
Description: as for outcome 6
Time Frame: At one month after Dose 2 of Havrix® vaccine (Month 8-11)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Prevnar Havrix Group
Number analyzed (Participants) | 115
mIU/mL | 1391.2 [1092.5 to 1771.4]

9. Secondary Outcome: Number of Subjects With Vaccine Response to Anti-HAV Antibodies
Description: The vaccine response was defined as:
  1. a detectable anti-HAV antibody concentration one month after Dose 2 in subjects who were initially seronegative (antibody concentrations < 15 mIU/mL for anti-HAV); or
  2. a 2-fold increase above the pre-vaccination concentration one month after Dose 2 in subjects who were initially seropositive (antibody concentrations ≥ 15 mIU/mL for anti-HAV).
Time Frame: One month after Dose 2 of Havrix® vaccine (Month 7-10/8-10)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Havrix Group | Havrix+Prevnar Group | Prevnar Havrix Group
Number analyzed (Participants) | 102 | 90 | 112
Participants | 102 | 89 | 110

10. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade. Grade 3 pain = cried when limb was moved/spontaneously painful. Grade 3 redness/swelling = redness/swelling spreading beyond 20 millimeters (mm) of injection site.
Time Frame: During the 4-day (Day 0-3) follow-up period after each vaccine dose and across doses
Population: The analysis was performed on the Total Vaccinated Cohort, which included all vaccinated subjects with at least one study vaccine administration documented and with the symptoms sheet filled in.
Measure: Count of Participants; unit: Participants
Arm/Group | Havrix Group | Havrix+Prevnar Group | Prevnar Havrix Group
Number analyzed (Participants) | 141 | 133 | 142
Participants
  Any Pain, Dose 1: number analyzed (Participants) | 139 | 133 | 140
  Any Pain, Dose 1 | 39 | 48 | 61
  Grade 3 Pain, Dose 1: number analyzed (Participants) | 139 | 133 | 140
  Grade 3 Pain, Dose 1 | 0 | 2 | 1
  Any Redness, Dose 1: number analyzed (Participants) | 139 | 133 | 140
  Any Redness, Dose 1 | 31 | 54 | 64
  Grade 3 Redness, Dose 1: number analyzed (Participants) | 139 | 133 | 140
  Grade 3 Redness, Dose 1 | 0 | 7 | 7
  Any Swelling, Dose 1: number analyzed (Participants) | 139 | 133 | 140
  Any Swelling, Dose 1 | 9 | 39 | 38
  Grade 3 Swelling, Dose 1: number analyzed (Participants) | 139 | 133 | 140
  Grade 3 Swelling, Dose 1 | 0 | 5 | 2
  Any Pain, Dose 2: number analyzed (Participants) | 123 | 114 | 130
  Any Pain, Dose 2 | 34 | 34 | 35
  Grade 3 Pain, Dose 2: number analyzed (Participants) | 123 | 114 | 130
  Grade 3 Pain, Dose 2 | 0 | 1 | 1
  Any Redness, Dose 2: number analyzed (Participants) | 123 | 114 | 130
  Any Redness, Dose 2 | 30 | 28 | 37
  Grade 3 Redness, Dose 2: number analyzed (Participants) | 123 | 114 | 130
  Grade 3 Redness, Dose 2 | 0 | 1 | 0
  Any Swelling, Dose 2: number analyzed (Participants) | 123 | 114 | 130
  Any Swelling, Dose 2 | 12 | 18 | 17
  Grade 3 Swelling, Dose 2: number analyzed (Participants) | 123 | 114 | 130
  Grade 3 Swelling, Dose 2 | 0 | 1 | 0
  Any Pain, Dose 3: number analyzed (Participants) | 141 | 133 | 127
  Any Pain, Dose 3 | NA — No Dose 3 was administered to this group. | NA — No Dose 3 was administered to this group. | 29
  Grade 3 Pain, Dose 3: number analyzed (Participants) | 141 | 133 | 127
  Grade 3 Pain, Dose 3 | NA — No Dose 3 was administered to this group. | NA — No Dose 3 was administered to this group. | 0
  Any Redness, Dose 3: number analyzed (Participants) | 141 | 133 | 127
  Any Redness, Dose 3 | NA — No Dose 3 was administered to this group. | NA — No Dose 3 was administered to this group. | 32
  Grade 3 Redness, Dose 3: number analyzed (Participants) | 141 | 133 | 127
  Grade 3 Redness, Dose 3 | NA — No Dose 3 was administered to this group. | NA — No Dose 3 was administered to this group. | 0
  Any Swelling, Dose 3: number analyzed (Participants) | 141 | 133 | 127
  Any Swelling, Dose 3 | NA — No Dose 3 was administered to this group. | NA — No Dose 3 was administered to this group. | 16
  Grade 3 Swelling, Dose 3: number analyzed (Participants) | 141 | 133 | 127
  Grade 3 Swelling, Dose 3 | NA — No Dose 3 was administered to this group. | NA — No Dose 3 was administered to this group. | 0
  Any Pain, Across Doses | 57 | 62 | 76
  Grade 3 Pain, Across Doses | 0 | 3 | 2
  Any Redness, Across Doses | 45 | 64 | 78
  Grade 3 Redness, Across Doses | 0 | 8 | 7
  Any Swelling, Across Doses | 19 | 47 | 48
  Grade 3 Swelling, Across Doses | 0 | 6 | 2

11. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms
Description: Assessed solicited general symptoms were drowsiness, fever [defined as axillary temperature equal to or above (≥) 37.5 degrees Celsius (°C)], irritability and loss of appetite. Any = occurrence of the symptom regardless of intensity grade. Grade 3 drowsiness = drowsiness that prevented normal activity. Grade 3 fever = fever > 39.0 °C. Grade 3 irritability = crying that could not be comforted/prevented normal activity. Grade 3 loss of appetite = not eating at all. Related = symptom assessed by the investigator as related to the vaccination.
Time Frame: During the 4-day (Day 0-3) follow-up period after each vaccine dose and across doses
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Havrix Group | Havrix+Prevnar Group | Prevnar Havrix Group
Number analyzed (Participants) | 141 | 133 | 142
Participants
  Any Drowsiness, Dose 1: number analyzed (Participants) | 139 | 133 | 140
  Any Drowsiness, Dose 1 | 40 | 35 | 45
  Grade 3 Drowsiness, Dose 1: number analyzed (Participants) | 139 | 133 | 140
  Grade 3 Drowsiness, Dose 1 | 2 | 2 | 3
  Related Drowsiness, Dose 1: number analyzed (Participants) | 139 | 133 | 140
  Related Drowsiness, Dose 1 | 34 | 34 | 39
  Any Fever, Dose 1: number analyzed (Participants) | 139 | 133 | 140
  Any Fever, Dose 1 | 12 | 19 | 23
  Grade 3 Fever, Dose 1: number analyzed (Participants) | 139 | 133 | 140
  Grade 3 Fever, Dose 1 | 0 | 1 | 2
  Related Fever, Dose 1: number analyzed (Participants) | 139 | 133 | 140
  Related Fever, Dose 1 | 11 | 11 | 18
  Any Irritability, Dose 1: number analyzed (Participants) | 139 | 133 | 140
  Any Irritability, Dose 1 | 48 | 47 | 58
  Grade 3 Irritability, Dose 1: number analyzed (Participants) | 139 | 133 | 140
  Grade 3 Irritability, Dose 1 | 0 | 0 | 2
  Related Irritability, Dose 1: number analyzed (Participants) | 139 | 133 | 140
  Related Irritability, Dose 1 | 44 | 44 | 50
  Any Loss of appetite, Dose 1: number analyzed (Participants) | 139 | 133 | 140
  Any Loss of appetite, Dose 1 | 36 | 33 | 35
  Grade 3 Loss of appetite, Dose 1: number analyzed (Participants) | 139 | 133 | 140
  Grade 3 Loss of appetite, Dose 1 | 1 | 2 | 2
  Related Loss of appetite, Dose 1: number analyzed (Participants) | 139 | 133 | 140
  Related Loss of appetite, Dose 1 | 31 | 24 | 27
  Any Drowsiness, Dose 2: number analyzed (Participants) | 123 | 116 | 129
  Any Drowsiness, Dose 2 | 18 | 27 | 28
  Grade 3 Drowsiness, Dose 2: number analyzed (Participants) | 123 | 116 | 129
  Grade 3 Drowsiness, Dose 2 | 0 | 2 | 0
  Related Drowsiness, Dose 2: number analyzed (Participants) | 123 | 116 | 129
  Related Drowsiness, Dose 2 | 16 | 25 | 25
  Any Fever, Dose 2: number analyzed (Participants) | 123 | 116 | 129
  Any Fever, Dose 2 | 12 | 7 | 10
  Grade 3 Fever, Dose 2: number analyzed (Participants) | 123 | 116 | 129
  Grade 3 Fever, Dose 2 | 1 | 1 | 2
  Related Fever, Dose 2: number analyzed (Participants) | 123 | 116 | 129
  Related Fever, Dose 2 | 12 | 6 | 7
  Any Irritability, Dose 2: number analyzed (Participants) | 123 | 116 | 129
  Any Irritability, Dose 2 | 28 | 36 | 42
  Grade 3 Irritability, Dose 2: number analyzed (Participants) | 123 | 116 | 129
  Grade 3 Irritability, Dose 2 | 1 | 0 | 1
  Related Irritability, Dose 2: number analyzed (Participants) | 123 | 116 | 129
  Related Irritability, Dose 2 | 26 | 34 | 40
  Any Loss of appetite, Dose 2: number analyzed (Participants) | 123 | 116 | 129
  Any Loss of appetite, Dose 2 | 15 | 20 | 24
  Grade 3 Loss of appetite, Dose 2: number analyzed (Participants) | 123 | 116 | 129
  Grade 3 Loss of appetite, Dose 2 | 1 | 2 | 0
  Related Loss of appetite, Dose 2: number analyzed (Participants) | 123 | 116 | 129
  Related Loss of appetite, Dose 2 | 14 | 17 | 21
  Any Drowsiness, Dose 3: number analyzed (Participants) | 141 | 133 | 129
  Any Drowsiness, Dose 3 | NA — No Dose 3 was administered to this group. | NA — No Dose 3 was administered to this group. | 20
  Grade 3 Drowsiness, Dose 3: number analyzed (Participants) | 141 | 133 | 129
  Grade 3 Drowsiness, Dose 3 | NA — No Dose 3 was administered to this group. | NA — No Dose 3 was administered to this group. | 0
  Related Drowsiness, Dose 3: number analyzed (Participants) | 141 | 133 | 129
  Related Drowsiness, Dose 3 | NA — No Dose 3 was administered to this group. | NA — No Dose 3 was administered to this group. | 18
  Any Fever, Dose 3: number analyzed (Participants) | 141 | 133 | 129
  Any Fever, Dose 3 | NA — No Dose 3 was administered to this group. | NA — No Dose 3 was administered to this group. | 10
  Grade 3 Fever, Dose 3: number analyzed (Participants) | 141 | 133 | 129
  Grade 3 Fever, Dose 3 | NA — No Dose 3 was administered to this group. | NA — No Dose 3 was administered to this group. | 1
  Related Fever, Dose 3: number analyzed (Participants) | 141 | 133 | 129
  Related Fever, Dose 3 | NA — No Dose 3 was administered to this group. | NA — No Dose 3 was administered to this group. | 9
  Any Irritability, Dose 3: number analyzed (Participants) | 141 | 133 | 129
  Any Irritability, Dose 3 | NA — No Dose 3 was administered to this group. | NA — No Dose 3 was administered to this group. | 27
  Grade 3 Irritability, Dose 3: number analyzed (Participants) | 141 | 133 | 129
  Grade 3 Irritability, Dose 3 | NA — No Dose 3 was administered to this group. | NA — No Dose 3 was administered to this group. | 0
  Related Irritability, Dose 3: number analyzed (Participants) | 141 | 133 | 129
  Related Irritability, Dose 3 | NA — No Dose 3 was administered to this group. | NA — No Dose 3 was administered to this group. | 27
  Any Loss of appetite, Dose 3: number analyzed (Participants) | 141 | 133 | 129
  Any Loss of appetite, Dose 3 | NA — No Dose 3 was administered to this group. | NA — No Dose 3 was administered to this group. | 16
  Grade 3 Loss of appetite, Dose 3: number analyzed (Participants) | 141 | 133 | 129
  Grade 3 Loss of appetite, Dose 3 | NA — No Dose 3 was administered to this group. | NA — No Dose 3 was administered to this group. | 1
  Related Loss of appetite, Dose 3: number analyzed (Participants) | 141 | 133 | 129
  Related Loss of appetite, Dose 3 | NA — No Dose 3 was administered to this group. | NA — No Dose 3 was administered to this group. | 14
  Any Drowsiness, Across | 48 | 49 | 63
  Grade 3 Drowsiness, Across | 2 | 4 | 6
  Related Drowsiness, Across | 41 | 47 | 58
  Any Fever, Across | 21 | 24 | 31
  Grade 3 Fever, Across | 1 | 2 | 4
  Related Fever, Across | 20 | 17 | 26
  Any Irritability, Across | 60 | 65 | 82
  Grade 3 Irritability, Across | 1 | 0 | 3
  Related Irritability, Across | 55 | 63 | 79
  Any Loss of appetite, Across | 42 | 45 | 54
  Grade 3 Loss of appetite, Across | 2 | 4 | 3
  Related Loss of appetite, Across | 37 | 36 | 49

12. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Unsolicited Adverse Events (AEs)
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination. Grade 3 AE = an AE which prevented normal, everyday activities. Related = AE assessed by the investigator as related to the vaccination.
Time Frame: During the 31-day (Day 0-30) follow-up period
Population: The analysis was performed on the Total Vaccinated Cohort, which included all vaccinated subjects with at least one study vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | Havrix Group | Havrix+Prevnar Group | Prevnar Havrix Group
Number analyzed (Participants) | 147 | 137 | 149
Participants
  Any AE(s) | 82 | 72 | 87
  Grade 3 AE(s) | 3 | 5 | 8
  Related AE(s) | 8 | 8 | 12

13. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs), New Chronic Illnesses (NCIs) and Medically Significant Events (MSEs)
Description: SAEs assessed include medical occurrences that result in death, are life-threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity. NCIs include autoimmune disorders, asthma, type I diabetes, allergies. MSEs include AEs prompting emergency room or physician visits that are not related to common diseases or routine visits for physical examination or vaccination, or serious adverse events (SAEs) that are not related to common diseases. Common diseases include upper respiratory infections, sinusitis, pharyngitis, gastroenteritis, urinary tract infections, cervico-vaginal yeast infections, menstrual cycle abnormalities and injury.
Time Frame: During the Active Phase (from Day 0 to Day 30 after final vaccine dose for each subject)
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Havrix Group | Havrix+Prevnar Group | Prevnar Havrix Group
Number analyzed (Participants) | 147 | 137 | 149
Participants
  Any SAE(s) | 3 | 5 | 5
  Any NCI(s) | NA — New chronic illnesses were only collected in the Extended Safety Follow-up (ESFU) Phase, therefore all the unsolicited AEs throughout the study were reported without identifying which AEs were considered a new chronic illness. | NA — New chronic illnesses were only collected in the Extended Safety Follow-up (ESFU) Phase, therefore all the unsolicited AEs throughout the study were reported without identifying which AEs were considered a new chronic illness. | NA — New chronic illnesses were only collected in the Extended Safety Follow-up (ESFU) Phase, therefore all the unsolicited AEs throughout the study were reported without identifying which AEs were considered a new chronic illness.
  Any MSE(s) | NA — Related information about medically significant events was not specifically collected in the Case Report Form, therefore, all the unsolicited AEs throughout the study were reported without identifying which AEs were considered medically significant. | NA — Related information about medically significant events was not specifically collected in the Case Report Form, therefore, all the unsolicited AEs throughout the study were reported without identifying which AEs were considered medically significant. | NA — Related information about medically significant events was not specifically collected in the Case Report Form, therefore, all the unsolicited AEs throughout the study were reported without identifying which AEs were considered medically significant.

14. Secondary Outcome: Number of Subjects With SAEs, NCIs and MSEs
Description: SAEs assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity. NCIs include autoimmune disorders, asthma, type I diabetes, allergies. MSEs include AEs prompting emergency room or physician visits that are not related to common diseases or routine visits for physical examination or vaccination, or serious adverse events (SAEs) that are not related to common diseases. Common diseases include upper respiratory infections, sinusitis, pharyngitis, gastroenteritis, urinary tract infections, cervico-vaginal yeast infections, menstrual cycle abnormalities and injury.
Time Frame: During the Extended Safety Follow-up (ESFU) Phase (from Day 30 to 6 months after final vaccine dose)
Population: The analysis was performed on the ESFU cohort, which included all vaccinated subjects for whom safety data were available during the extended safety follow-up period (from Day 30 up to 6 months after last vaccine dose).
Measure: Count of Participants; unit: Participants
Arm/Group | Havrix Group | Havrix+Prevnar Group | Prevnar Havrix Group
Number analyzed (Participants) | 123 | 121 | 132
Participants
  Any SAE(s) | 0 | 2 | 3
  Any NCI(s) | NA — All the unsolicited AEs throughout the study were reported without identifying which AEs were considered a new chronic illness. | NA — All the unsolicited AEs throughout the study were reported without identifying which AEs were considered a new chronic illness. | NA — All the unsolicited AEs throughout the study were reported without identifying which AEs were considered a new chronic illness.
  Any MSE(s) | NA — All the unsolicited AEs throughout the study were reported without identifying which AEs were considered medically significant. | NA — All the unsolicited AEs throughout the study were reported without identifying which AEs were considered medically significant. | NA — All the unsolicited AEs throughout the study were reported without identifying which AEs were considered medically significant.

ADVERSE EVENTS:
Time Frame: Solicited local and general AEs: during the 4-day (Day 0-3); Unsolicited AEs: during the 31-day (Day 0-30); SAEs, NCIs and MSEs: during the entire study period(from Month 0 to Month 12-15/13-16).
Arm/Group | Havrix Group | Havrix+Prevnar Group | Prevnar Havrix Group
Serious Adverse Events (participants affected / at risk) | 6/177 | 8/169 | 10/175
Other Adverse Events (participants affected / at risk) | 107/147 | 106/137 | 121/149
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Havrix Group (N=177) | Havrix+Prevnar Group (N=169) | Prevnar Havrix Group (N=175)
Bronchiolitis (enrollment phase) (Infections and infestations) | 1 | 0 | 0
Burns second degree (enrolllment phase) (Injury, poisoning and procedural complications) | 0 | 0 | 1
Convulsion (enrollment phase) (Nervous system disorders) | 1 | 1 | 0
Gastroenteritis (enrollment phase) (Infections and infestations) | 1 | 0 | 0
Lactose intolerance (enrollment phase) (Metabolism and nutrition disorders) | 0 | 0 | 1
Otitis media acute (enrollment phase) (Infections and infestations) | 2 | 0 | 0
Upper respiratory tract infection (enrollment phase) (Infections and infestations) | 1 | 0 | 0
Convulsion (active phase) (Nervous system disorders) | 1/147 | 0/137 | 1/149
Croup infectious (active phase) (Infections and infestations) | 1/147 | 1/137 | 0/149
Pneumonia (active phase) (Infections and infestations) | 0/147 | 2/137 | 0/149
Bronchial hyperactivity (active phase) (Respiratory, thoracic and mediastinal disorders) | 0/147 | 0/137 | 1/149
Bronchiolitis (active phase) (Infections and infestations) | 0/147 | 0/137 | 1/149
Dehydration (active phase) (Metabolism and nutrition disorders) | 0/147 | 1/137 | 0/149
Developmental delay (active phase) (General disorders) | 0/147 | 1/137 | 0/149
Diabetes mellitus insulin-dependent (active phase) (Metabolism and nutrition disorders) | 0/147 | 0/137 | 1/149
Gait disturbance (active phase) (General disorders) | 0/147 | 1/137 | 0/149
Gastroenteritis viral (Infections and infestations) | 0/147 | 0/137 | 1/149
Hearing impaired (active phase) (Ear and labyrinth disorders) | 0/147 | 1/137 | 0/149
Hypoxia (active phase) (Respiratory, thoracic and mediastinal disorders) | 0/147 | 1/137 | 0/149
Kawasaki's disease (active phase) (Infections and infestations) | 1/147 | 0/137 | 0/149
Langerhans' cell granulomatosis (active phase) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/147 | 1/137 | 0/149
Dehydration (ESFU phase) (Metabolism and nutrition disorders) | 0/123 | 0/121 | 2/132
Gastroenteritis viral (ESFU phase) (Infections and infestations) | 0/123 | 1/121 | 1/132
Kawasaki's disease (ESFU phase) (Infections and infestations) | 0/123 | 0/121 | 1/132
Pneumonia (ESFU phase) (Infections and infestations) | 0/123 | 1/121 | 0/132
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Havrix Group (N=147) | Havrix+Prevnar Group (N=137) | Prevnar Havrix Group (N=149)
Pain (General disorders) | 57/141 | 62/133 | 76/142
Redness (General disorders) | 45/141 | 64/133 | 78/142
Swelling (General disorders) | 19/141 | 47/133 | 48/142
Drowsiness (General disorders) | 48/141 | 49/133 | 63/142
Fever (Axillary) (General disorders) | 21/141 | 24/133 | 31/142
Irritability (General disorders) | 60/141 | 65/133 | 82/142
Loss of appetite (General disorders) | 42/141 | 45/133 | 54/142
Upper respiratory tract infection (Infections and infestations) | 22 | 17 | 26
Otitis media (Infections and infestations) | 14 | 20 | 27
Pyrexia (General disorders) | 10 | 8 | 12
Diarrhea (Gastrointestinal disorders) | 8 | 8 | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 5 | 8
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 13

LIMITATIONS AND CAVEATS:
None reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.